CLINICAL TRIAL: NCT02261025
Title: The Effect Of Aspirin On Survival in in Patients Undergoing Chronic Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hui Min Jin, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20120308
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Hemodialysis
Keywords: aspirin
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin group (Experimental): Aspirin 75-100mg,per day，oral
  Interventions: Drug: acetylsalicylic acid
- non-aspirin group (No Intervention): No interventions

INTERVENTIONS:
Drug: acetylsalicylic acid — 75-100mg,per day
  Other Names: Aspirin
  Arms: Aspirin group

SUMMARY:
The aim of present study is to examine the effect of low-dose aspirin on the incidence of cardiovascular events and mortality in patients undergoing chronic hemodialysis.

DETAILED DESCRIPTION:
This study prospectively evaluate the impacts of low dose aspirin on survival and cardio-cerebral vascular events in a large cohort of Chinese patients undergoing chronic hemodialysis. Between January 2008, consecutive patients with hemodialysis with aspirin were enrolled.We examine the association of aspirin with all-cause mortality in patients matched by propensity scores using the Kaplan-Meier method and Cox models in "intention-to-treat" analyses.The secondary endpoint was rate of cardio-cerebral events.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 18 to 85, undergoing chronic hemodialysis, who have none of the following exclusion criteria.

Exclusion Criteria:

History of gastric or duodenal ulcers Known allergy to aspirin or other NSAIDs

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2008-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
survival rate | 5 years

SECONDARY OUTCOMES:
cardio-cerebral event | 5 years

REFERENCES:
- [Derived] Liu J, Pan Y, Chen L, Qiao QY, Wang J, Pan LH, Gu YH, Gu HF, Fu SK, Jin HM. Low-dose aspirin for prevention of cardiovascular disease in patients on hemodialysis: A 5-y prospective cohort study. Hemodial Int. 2016 Oct;20(4):548-557. doi: 10.1111/hdi.12409. Epub 2016 Mar 1. PMID 26932276